CLINICAL TRIAL: NCT03358511
Title: Engineering Gut Microbiome to Target Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Saranya Chumsri, Associate Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-002215
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast Cancer Patients (Experimental): All subjects will be given 2-4 weeks of probiotics prior to surgery in operable stage I-III breast adenocarcinoma tumors ≥1.0 cm. Subjects will take the probiotic three times a day.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Primal Defense Ultra® Probiotic Formula is an over-the-counter probiotic that provides 15 billion colony forming units of 13 species of beneficial bacteria, including Saccharomyces boulardii, Lactobacillus plantarum, Bacillus subtilis, Bifidobacterium lactis, Bifidobacterium bifidum, Lactobacillus rhamnosus, Bifidobacterium breve, lactobacillus casei, Lactobacillus salivarius, Lactobacillus acidophilus, Lactobacillus brevis, Bifidobacterium longum, and Lactobacillus paracasei.
  Other Names: Primal Defense ULTRA Probiotic Formula

SUMMARY:
The purpose of this study is to find out if using probiotics will help the body's immune system react to breast cancer. New studies showed that diverse species of bacteria inside the bowel might help improve immune system, particularly the ability of immune system to recognize cancer. This study will investigate how probiotics will affect the subjects' immune system on breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females ≥ 18 years of age
* Histologically confirmed adenocarcinoma of the breast ≥1.0 cm operable stage I-III
* Must have adequate organ function,
* Not receive systemic neoadjuvant therapy
* Be willing to provide tissue, blood, and stool samples for research study.
* Must not have taken any probiotics in the past 60 days prior to enrollment.

Exclusion Criteria:

* Patients with autoimmune disease, immune deficiency such as HIV, irritable bowel, known diverticulosis, and other serious GI conditions at treating physician's discretion will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Mean number of cytotoxic T lymphocytes (CD8+ cells) | Approximately 4 weeks after baseline
  CD8+ T cells (often called cytotoxic T lymphocytes) are very important for immune defence against intracellular pathogens, including viruses and bacteria, and for tumor surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials